CLINICAL TRIAL: NCT03939611
Title: The Effect of Foot Reflexology on Infantile Colic Symptoms: Randomized, Placebo-Controlled Trial
Brief Title: The Effect of Foot Reflexology on Infantile Colic Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, NIMET KARATAS, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AkdenizUniversity
Record Dates: First submitted 2019-05-02; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Infantile Colic; Reflexology
Keywords: complementary therapies; infantile colic; nurses; reflexology
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: This was an experimental, single-blind, randomized, placebo-controlled trial.
Who Masked: Participant
Masking Description: All parents were only told that foot application would be done, without giving any expectations. In the statistical analysis, the groups were named Group-1 and Group-2, and the statistician was blinded when evaluating the outputs. The report was written by the statistician, who did not know which application was performed to which group blinding was provided in the report writing. The scales were evaluated by the researcher, who could not be blinded due to the nature of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot Reflexology Group (Experimental): Foot reflexology was performed to the reflexology group infants. Foot reflexology application (FRA) involved relaxation for the first 3-5 minutes and the last 2 minutes; the remaining 12-15 minutes included stimulation of the brain and digestive system organs. To ensure relaxation, rotation was performed by using the thumbs of the hand under the feet, cephalocaudally. The session of FRA included stimulating the brain and medulla spinalis (2 min), the solar plexus (1min), the stomach (2min), the liver (2min), the pancreas (2min), the gallbladder (1min), and the ileocecal valve and intestine (5min) reflex points. Application was performed on all infants twice a week, for a total of four times during two consecutive weeks. Between two consecutive applications, a minimum of 48 hours and a maximum of 5 days was allotted (Stone, 2011). A total of 6 follow-ups were performed during the study period.
  Interventions: Other: Foot Reflexology
- Placebo Foot Reflexology Group (Placebo Comparator): Placebo foot reflexology was performed to the placebo group infants. Placebo foot reflexology application (PFRA) was constrained to ineffective touch without any stimulation and pressure. The aim of the PFRA was to create only a touch effect. It was applied by patted the foot by using the thumbs of the hand, for 20 minutes with the same rotation and to the same points as FRA. Application was performed on all infants twice a week, for a total of four times during two consecutive weeks. Between two consecutive applications, a minimum of 48 hours and a maximum of 5 days was allotted (Stone, 2011). A total of 6 follow-ups were performed during the study period.
  Interventions: Other: Placebo Foot Reflexology

INTERVENTIONS:
Other: Foot Reflexology — Reflexology is one of the complementary health approaches; it is based on systematic pressure and stimulation with fingers to energy points in feet and hands and is a topic nowadays studied. Reflexology argues that the reflex maps in the hands and feet with all of the parts of the body are in contact. The pressure applied to each point stimulates the circulation of blood and energy like a sensor, gives a sense of relaxation, provides homeostasis. With a touch that is a different way of communication with children, is supported to create physical awareness via reflexology techniques, and is provided healthy nutrition of the stimulated tissue.
  Arms: Foot Reflexology Group
Other: Placebo Foot Reflexology — Placebo reflexology was performed by touch without pressure to the same rotation and to the same points as foot reflexology application. It was performed only to compare foot reflexology with a placebo effect.
  Arms: Placebo Foot Reflexology Group

SUMMARY:
Aim: To compare the effect of foot reflexology and placebo foot reflexology on colic symptoms such as pain, ineffective sleep, and colicky crying periods in infants with colic.

Method: The study was conducted as a single-blind, randomized, placebo-controlled trial in a child hospital between June 2016 and March 2017. To start with, 20 infants with colic were randomly selected for the reflexology group, and 25 babies with colic were randomly selected for the placebo group. Simple randomization was used; the parents and statistician were blinded to group assessment. The researcher could not be blinded because of the role played in the study. Foot reflexology was implemented with reflexology-group infants. Placebo foot reflexology was used with placebo-group infants. Both interventions were performed four times, for 20 minutes, each, by the researcher over the course of two weeks. The data were collected by the researcher using the information form, infantile colic scale, behavioral pain scale, crying and sleeping follow-up forms.

ELIGIBILITY:
Inclusion Criteria:

Infants were included who were aged 1-3 months, Infants who were diagnosed IC by a pediatrician according to Wessel's rule of threes.

Exclusion Criteria (Beckmann & Le Quesne, 2005):

Infants who were using any of analgesic drug until 3 hours before the applications and antibiotic or steroid due to treating an illness, Infants who had an acute fever, musculoskeletal disease, active shingles or infection, acute shingles, or tissue in the foot and joint, All infants with any non-IC health problems.

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2016-06-26 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Infantile Colic State | In two weeks
  Ellet et al. (2002) developed a Likert-type scale to determine the factors causing colic and to diagnose colic. The scale consists of 5 sub-dimensions and 22 items. Sub-dimensions include 'Cow's Milk/Soy Protein Allergy/Intolerance', 'Immature Gastrointestinal System', 'Immature Central Nervous System', 'Difficult Infant Temperament', and 'Parent-Infant Interaction + Problem Infant'. These headings include factors affecting the infant's colic, such as sleep characteristics, consolability, features of crying, infant mood, and parent-infant interaction. The Cronbach's α coefficient of the scale was .69 (Ellett et al., 2003). Cetinkaya and Başbakkal (2007) tested the validity and reliability of the scale for the Turkish population and reported Cronbach's α to be .73 (Cetinkaya & Basbakkal, 2007). In this study, it was determined to be .65.
Colicky Pain | In two weeks
  The FLACC scale developed by Merkel et al. in 1997 is used to help determine the level of pain in infants and children. The parameters of scale include infant 'Facial expressions, Leg movements, Activities, Crying, and Consolability' (Voepel-Lewis, Shayevitz, & Malviya, 1997). The maximum score of this scale is ten, shows the highest pain. On the other hands; the minimum score is zero, shows that no pain. Şenaylı et al. (2006) reported that the scale could be used in Turkish population (Şenaylı, Özkan, Şenaylı, & Bıçakçı, 2006).
Colicky Crying | In two weeks
  Crying follow-up form was prepared by the researcher to determine the duration of crying in infants. Colic crying differs from ordinary crying as it is louder than normal and inconsolable. It occurs usually suddenly and takes several consecutive hours (Helseth, 2002). Based on this information, when crying ended, parents were asked to record crying times over half an hour, with start and end times. The form required hourly recording by the parents for two weeks.

SECONDARY OUTCOMES:
Sleeping | In two weeks
  Sleeping follow-up form was prepared by the researcher to determine the duration of sleeping in infants. The form required hourly recording by the parents for two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül İŞLER DALGIÇ, Professor, Principal Investigator — Corresponding Author

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandrovich I, Rakovitskaya O, Kolmo E, Sidorova T, Shushunov S. The effect of fennel (Foeniculum Vulgare) seed oil emulsion in infantile colic: a randomized, placebo-controlled study. Altern Ther Health Med. 2003 Jul-Aug;9(4):58-61. PMID 12868253
- [Background] Bennedbaek O, Viktor J, Carlsen KS, Roed H, Vinding H, Lundbye-Christensen S. [Infants with colic. A heterogenous group possible to cure? Treatment by pediatric consultation followed by a study of the effect of zone therapy on incurable colic]. Ugeskr Laeger. 2001 Jul 2;163(27):3773-8. Danish. PMID 11466984
- [Background] Cetinkaya B, Basbakkal Z. A validity and reliability study investigating the Turkish version of the Infant Colic Scale. Gastroenterol Nurs. 2007 Mar-Apr;30(2):84-90; discussion 90. doi: 10.1097/01.SGA.0000267925.31803.30. PMID 17440307
- [Background] Chandrababu R, Rathinasamy EL, Suresh C, Ramesh J. Effectiveness of reflexology on anxiety of patients undergoing cardiovascular interventional procedures: A systematic review and meta-analysis of randomized controlled trials. J Adv Nurs. 2019 Jan;75(1):43-53. doi: 10.1111/jan.13822. Epub 2018 Sep 5. PMID 30109722
- [Background] Cirgin Ellett ML, Murphy D, Stroud L, Shelton RA, Sullivan A, Ellett SG, Ellett LD. Development and psychometric testing of the infant colic scale. Gastroenterol Nurs. 2003 May-Jun;26(3):96-103. doi: 10.1097/00001610-200305000-00002. PMID 12811319
- [Background] Embong NH, Soh YC, Ming LC, Wong TW. Revisiting reflexology: Concept, evidence, current practice, and practitioner training. J Tradit Complement Med. 2015 Sep 28;5(4):197-206. doi: 10.1016/j.jtcme.2015.08.008. eCollection 2015 Oct. PMID 26587391
- [Background] Cohen Engler A, Hadash A, Shehadeh N, Pillar G. Breastfeeding may improve nocturnal sleep and reduce infantile colic: potential role of breast milk melatonin. Eur J Pediatr. 2012 Apr;171(4):729-32. doi: 10.1007/s00431-011-1659-3. Epub 2011 Dec 29. PMID 22205210
- [Background] Helseth S. Help in times of crying: nurses' approach to parents with colicky infants. J Adv Nurs. 2002 Nov;40(3):267-74. doi: 10.1046/j.1365-2648.2002.02368.x. PMID 12383178
- [Background] Icke S, Genc R. Effect of Reflexology on Infantile Colic. J Altern Complement Med. 2018 Jun;24(6):584-588. doi: 10.1089/acm.2017.0315. Epub 2018 Apr 20. PMID 29676928
- [Background] Johnson JD, Cocker K, Chang E. Infantile Colic: Recognition and Treatment. Am Fam Physician. 2015 Oct 1;92(7):577-82. PMID 26447441
- [Background] Koc T, Gozen D. The Effect of Foot Reflexology on Acute Pain in Infants: A Randomized Controlled Trial. Worldviews Evid Based Nurs. 2015 Oct;12(5):289-96. doi: 10.1111/wvn.12099. Epub 2015 Jul 28. PMID 26220257
- [Background] Landgren K, Hallstrom I. Parents' experience of living with a baby with infantile colic--a phenomenological hermeneutic study. Scand J Caring Sci. 2011 Jun;25(2):317-24. doi: 10.1111/j.1471-6712.2010.00829.x. Epub 2010 Aug 18. PMID 20723153
- [Background] Reinthal M, Lund I, Ullman D, Lundeberg T. Gastrointestinal symptoms of infantile colic and their change after light needling of acupuncture: a case series study of 913 infants. Chin Med. 2011 Aug 11;6:28. doi: 10.1186/1749-8546-6-28. PMID 21835014
- [Background] Savino F, Ceratto S, De Marco A, Cordero di Montezemolo L. Looking for new treatments of Infantile Colic. Ital J Pediatr. 2014 Jun 5;40:53. doi: 10.1186/1824-7288-40-53. PMID 24898541
- [Background] Savino F, Quartieri A, De Marco A, Garro M, Amaretti A, Raimondi S, Simone M, Rossi M. Comparison of formula-fed infants with and without colic revealed significant differences in total bacteria, Enterobacteriaceae and faecal ammonia. Acta Paediatr. 2017 Apr;106(4):573-578. doi: 10.1111/apa.13642. Epub 2016 Nov 15. PMID 27763733
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] WESSEL MA, COBB JC, JACKSON EB, HARRIS GS Jr, DETWILER AC. Paroxysmal fussing in infancy, sometimes called colic. Pediatrics. 1954 Nov;14(5):421-35. No abstract available. PMID 13214956
- [Background] Zeevenhooven J, Browne PD, L'Hoir MP, de Weerth C, Benninga MA. Infant colic: mechanisms and management. Nat Rev Gastroenterol Hepatol. 2018 Aug;15(8):479-496. doi: 10.1038/s41575-018-0008-7. PMID 29760502